CLINICAL TRIAL: NCT03438006
Title: A Prospective, Multi-centre Post Marketing Surveillance (PMS) Cohort Study to Monitor the Safety of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV)-16/18 L1 VLP AS04 Vaccine in Female Chinese Subjects Aged Between 9 and 45 Years, When Administered According to the Prescribing Information (PI) as Per Routine Practice.
Brief Title: A Post Marketing Surveillance (PMS) Study to Monitor the Safety of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) Vaccine in Female Chinese Subjects
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207350
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Safety; Human Papillomavirus Vaccine; Adverse Event Following Immunization
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervarix group: Healthy female Chinese subjects aged between 9 and 45 years, vaccinated according to the Prescribing Information (PI) as per routine practice.
  Interventions: Other: Safety data collection (following routine vaccination)

INTERVENTIONS:
Other: Safety data collection (following routine vaccination) — This study assessed the safety of GSK Biologicals' Human papillomavirus (HPV) vaccine when administered routinely according to the Prescribing Information in female Chinese subjects aged between 9 and 45 years.
  The intervention consisted in the active surveillance of adverse events following immunization and pregnancy outcomes if the vaccine was administered inadvertently during pregnancy. Information of potential adverse events and pregnancy outcomes were collected at immunisation visits, telephone contacts and through spontaneous reporting by the patient/LAR/physician.

SUMMARY:
The purpose of this prospective, multi-centre, PMS cohort study was to monitor the safety of Cervarix, which is the first HPV vaccine licensed for use in China, to help prevent cervical cancer caused by HPV types 16 and 18. The vaccine was approved by National Drug Administration of China (CNDA), in July 2016.

As per the CNDA commitment, this study collected data regarding the safety of the vaccine, related information on potential immune-mediated diseases (pIMDs); which are diseases that could affect the immune system, and the effect on pregnancy outcomes (POs) including birth defects in the newborn.

Cervarix was approved for use in females between 9-25 years of age, for the prevention of cervical cancer, cervical intraepithelial neoplasia grade 1 (CIN1), cervical intraepithelial neoplasia grade 2, grade 3 (CIN 2/3) and adenocarcinoma in situ caused by high-risk human papillomavirus (HR-HPV) types 16 and 18.

In May 2018, Cervarix was also approved for use in women of age up to 45 years.

The exposed set (ES) comprised 3013 subjects, who were vaccinated with Cervarix, on a voluntary basis, as per standard practice. The study collected information on any adverse event following immunisation, pIMDs, POs and congenital anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Any Chinese female subject aged between 9 and 45 years, at the time of first vaccination dose, who received voluntary vaccination.
* Subjects for whom the investigator believed that they or their parent(s)/LAR(s) could and complied with the requirements mentioned in the protocol (e.g., return for the subsequent dose of vaccination and follow-up visits) were included in the study.
* Written informed consent was obtained from the subject. For subjects who were below the legal age of consent, written informed consent were obtained from the parent(s)/LAR(s) of the subject and informed assent were obtained from the subject according to EC requirement as well as local law.

Exclusion Criteria:

• Child in care

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy female Chinese subjects aged between 9 and 45 years, vaccinated on a voluntary basis as per standard practice.
Sampling Method: Non-Probability Sample
Enrollment: 3016 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- China (5):
  - GSK Investigational Site, Foshan, Guangdong
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Changzhou, Jiangsu
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Shanghai

REFERENCES:
- [Derived] Wu Q, Qian M, Welby S, Guignard A, Rosillon D, Gopala K, Xu Y, Liu K, He Y, Jiang N, Tan Q, Xie J, Zhu T, Wang Q, Pan Y, Zeng R, Yang J, Zhao X, Zhou M, Navarro-Torne A, Yu H, Borys D. Prospective, multi-center post-marketing surveillance cohort study to monitor the safety of the human papillomavirus-16/18 AS04-adjuvanted vaccine in Chinese girls and women aged 9 to 45 years, 2018-2020. Hum Vaccin Immunother. 2023 Dec 15;19(3):2283912. doi: 10.1080/21645515.2023.2283912. Epub 2023 Dec 1. PMID 38038626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centres in China
Pre-assignment Details: Out of 3016 participants enrolled in the study, 3 participants did not receive any vaccination and therefore were not included in any analysis.
Groups:
- Cervarix Group: Healthy female Chinese participants aged between 9 and 45 years, vaccinated according to the Prescribing Information (PI) as per routine practice.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 3013
Completed | 2895
Not Completed | 118
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 67
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 47
Not completed — NOT WILLING / NOT ABLE TO BE CONTACTED | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3013
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 30.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3013
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 3013

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any (Following Each Dose and Across Doses), Grade 3 (Across Doses) and Vaccine Related (Across Doses) Medically Attended Adverse Events Following Immunisation (AEFIs)
Description: An adverse event following immunisation (AEFI) is defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a vaccine. Medically attended AEFIs are defined as events leading to an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits. Any Medically attended AEFIS are presented for each dose and across doses. Grade 3 Medically attended AEFI = an AEFI which prevented normal, everyday activities. Related Medically Attended AEFI = AEFI assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day period following each immunisation with Cervarix (administered on Day 1, Month 1 and Month 6)
Population: Analysis was based on the Exposed Set (ES) which included all participants exposed to Cervarix and who provided safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3013
Participants
  Dose 1 | 49
  Dose 2: number analyzed (Participants) | 2956
  Dose 2 | 55
  Dose 3: number analyzed (Participants) | 2870
  Dose 3 | 56
  Across doses | 147
  Grade 3 | 1
  Related | 2

2. Secondary Outcome: Number of Participants With Any, Fatal and Vaccine Related Serious AEFIs (Across Doses)
Description: Serious AEFIs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a participant. Any serious AEFI = If a medically attended AEFI led to hospitalisation (or met any other serious AEFI criteria). Fatal Serious AEFIs are those events that resulted in death. Related Serious AEFIs= AEFIs assessed by the investigator as causally related to the study vaccination.
Time Frame: Throughout the study period (From Day 1 to either 12 months following the third immunisation (Month 18) or 24 months following the first immunisation with Cervarix (Month 24) whichever occured first))
Population: Analysis was based on the Exposed Set (ES) which included all participants exposed to Cervarix.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3013
Participants
  Any | 22
  Fatal | 0
  Related | 0

3. Secondary Outcome: Number of Participants With Any, Grade 3 and Vaccine Related Potential Immune Mediated Diseases (pIMDs) (Across Doses)
Description: pIMDs are a subset of AEFIs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which might or might not have an autoimmune aetiology. Any was defined as the occurrence of any pIMD regardless of intensity grade or relation to vaccination. Grade 3 pIMDs = pIMDs which prevented normal, everyday activities. Related pIMDs = pIMDs assessed by the investigator as related to the vaccination.
Time Frame: Throughout the study period (from Day 1 up to either 12 months following the third immunisation (Month 18) or 24 months following the first immunisation with Cervarix (Month 24), whichever occured first))
Population: Analysis was based on the Exposed Set (ES) which included all participants exposed to Cervarix.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 3013
Participants
  Any | 1
  Grade 3 | 0
  Related | 0

4. Secondary Outcome: Number of Participants Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: The number of participants reporting pregnancies and outcomes of reported pregnancies (elective abortion for medical reasons, spontaneous abortion or congenital anomaly) when Cervarix was administered to the participant, inadvertently within 60 days before pregnancy onset, or any time during pregnancy, was reported.
Time Frame: as for outcome 3
Population: The analysis was based on the ES, which included all participants exposed to Cervarix and who reported pregnancies and/or outcomes of reported pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 65
Participants
  Live infant no apparent congenital anomaly | 34
  Live infant congenital anomaly | 1
  Elective termination no apparent congenital anomaly | 20
  Elective termination congenital anomaly | 0
  Spontaneous abortion no apparent congenital anomaly | 1
  Spontaneous abortion congenital anomaly | 0
  Stillbirth no apparent congenital anomaly | 0
  Stillbirth congenital anomaly | 0
  Ectopic pregnancy | 4
  Molar pregnancy | 0
  Pregnancies lost to follow-up | 5
  Pregnancy ongoing | 0

ADVERSE EVENTS:
Time Frame: Medically attended Adverse Events Following Immunisation (AEFI): During 30-Days after each vaccination (administered on Day 1, Month 1 and Month 6). Serious AEFI: During the entire study period [starting at the first immunisation (Day 1) and ending either 12 months following the third immunisation (Month 18) or 24 months following the first immunisation with Cervarix (Month 24), whichever occured first].
Arm/Group | Cervarix Group
All-Cause Mortality (participants affected / at risk) | 0/3013
Serious Adverse Events (participants affected / at risk) | 22/3013
Other Adverse Events (participants affected / at risk) | 143/3013
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=3013)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Glycogen storage disease type I (Congenital, familial and genetic disorders) | 1 (1)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Mastitis (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Viral hepatitis carrier (Infections and infestations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1)
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Uterine scar (Reproductive system and breast disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 2 (2)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=3013)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Conjunctival oedema (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 4 (4)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 4 (5)
Pyrexia (General disorders) | 10 (10)
Hypersensitivity (Immune system disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 24 (26)
Conjunctivitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5)
Gingivitis (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 2 (2)
Herpangina (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Otitis media chronic (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 2 (2)
Periodontitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 9 (9)
Pneumonia (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 30 (32)
Urethritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5)
Vaginal infection (Infections and infestations) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 1 (1)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 3 (3)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT03438006/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03438006/SAP_001.pdf